CLINICAL TRIAL: NCT00956696
Title: Topiramate Treatment for Patients With Epilepsy and Learning Disability : A Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr Patrick Kwan, the Chinese University of Hong Kong
Other Study IDs: TPM2009
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Epilepsy
Keywords: Epilepsy; mental retardation
MeSH Terms: conditions — Epilepsy; Intellectual Disability | interventions — Topiramate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Topiramte: single arm, flexible dosing
  Interventions: Drug: topiramate

INTERVENTIONS:
Drug: topiramate — oral, daily dose or twice daily dose, total daily dose 25-200mg per day duration: 16 weeks
  Other Names: Topamax

SUMMARY:
It has been estimated that 22 - 32% of people with mental retardation or learning disability have co-existing epilepsy. Despite such high prevalence and although there may be particular concerns over the effects of treatment on behaviour and cognition in this population, few studies have specifically addressed these concerns. Topiramate (TPM) is one of the modern antiepileptic drugs that has been approved for the treatment of a broad range of seizure types in both children and adults. There is evidence of associated improvement in behaviour with treatment but data is conflicting. The investigators aim to further study the effect of TPM on seizure control and behaviour using the Scales of Independent Behavior-Revised (SIB-R) which has been applied in similar patient populations and is widely adopted locally to assess the behaviour of people with mental retardation. This is a naturalistic, open label, single arm prospective study of 16-week in duration. Eligible adult patients will be initiated on TPM. Patients will be evaluated at baseline, end of weeks 4, 10 and 16. At each visit seizure control and any adverse events will be assessed. Behaviour will be assessed using SIB-R (Chinese version) at baseline and each study visit. At the end of the study period the patient's overall improvement will be rated by the investigator and the caregiver using global evaluation scales. Patients with improvement will be maintained on TPM after the end of the study period Titration schedule Topiramate will be administered orally as per usual clinical practice. Treatment will be initiated at 25 mg daily for 1 week, and increased in 25- to 50-mg increments at one- to two-weekly intervals, to an initial target dose of 100 - 200 mg daily in 2 divided doses according to each individual's response. Further dose adjustment can be made in response to further seizures or emergence of adverse events..

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Patients mental retardation and with newly diagnosed epilepsy requiring treatment, or with chronic epilepsy that is unsatisfactorily controlled (defined as at least 2 seizures during an 8-week retrospective baseline).

Exclusion Criteria:

* History of nephrolithiasis or renal impairment
* Patients with absence seizures only
* History of status epilepticus in the previous 3 months while receiving appropriate antiepileptic drug therapy
* History of suicidal attempts or psychotic illness, psychiatric or mood disorders in the previous 6 months that required hospitalisation
* History of alcohol or drug abuse in the previous year
* Patients with progressive neurological conditions or terminal medical conditions.
* Patients whose seizures are thought to be of alcoholic, metabolic, neoplastic, infectious, or non-epileptic in origin (including psychogenic seizures).
* Chronic use of antacids, calcium supplements or high dose vitamin C.
* Women who are pregnant, lactating or without adequate contraception if they have child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Epilepsy patients in Prince of Wales hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Median monthly seizure frequency | 16 weeks

SECONDARY OUTCOMES:
Responder rate | 16 weeks
SIB-R score | 16 weeks
Investigator's global evaluation scale | 16 weeks
Caregivers' global evaluation scale | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kwan, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong